CLINICAL TRIAL: NCT02216110
Title: Long-term Outcomes of Endoscopic Submucosal Dissection Versus Gastrectomy for Early Gastric Cancer
Brief Title: Endoscopic Submucosal Dissection Versus Gastrectomy
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Assistant Professor, Soonchunhyang University Hospital
Other Study IDs: SCHDDC-2014-01
Record Dates: First submitted 2014-08-09; First posted 2014-08-13 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Early Gastric Cancer
Keywords: Endoscopic submucosal dissection; Gastrectomy; Survival; Outcome
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surgery group: Patients who underwent surgery as treatment of early gastric cancer
  Interventions: Procedure: Surgery
- ESD group: Patients who underwent endoscopic submucosal dissection (ESD) as treatment of early gastric cancer, instead of surgery

INTERVENTIONS:
Procedure: Surgery — Surgery for early gastric cancer includes distal gastrectomy, total gastrectomy, proximal gastrectomy, and wedge resection
  Groups: Surgery group

SUMMARY:
Gastrectomy is curative treatment for early gastric cancer (EGC). Recently, endoscopic submucosal dissection (ESD) has been accepted as standard treatment in selected patients with negligible risk of lymph node metastasis. However, there are limited data regarding the long-term outcomes of ESD in comparison with surgery. This protocol aims to compare overall survival rate, tumor recurrence, development of metachronous cancers after ESD and surgery.

DETAILED DESCRIPTION:
The prevalence of gastric cancer is high in Asia, especially in Korea and Japan. In Korea, the detection rate of EGC has increased with mass screening for the prevention of gastric cancer-related death. EGC is defined as mucosal or submucosal cancer, regardless of regional lymph node metastasis. The presence of lymph node metastasis has been reported to range from 2% to 18%. For this reason, radical gastrectomy with lymph node dissection was considered as the only curative treatment. In EGC patients, surgical outcome demonstrated excellent 5-year survival rate above 90%.

In 2000, EGC subgroups with negligible risk of lymph node metastasis were proposed on the basis of large scale retrospective data. Thereafter, the result was adopted as expanded criteria for endoscopic resection of EGC. ESD is useful technique to dissect the tumor along the submucosal layer using various endoscopic knives. Compared to endoscopic mucosal resection (EMR), ESD achieved a higher complete resection rate and a lower local tumor recurrence rate.

Although curative resection is pathologically achieved by ESD, post-resection surveillance is needed to confirm the presence of nodal metastasis. Recently, several studies reported that 5-year overall and disease-specific survival rate were highly favorable in EGC patients who underwent curative ESD. However, there is no comparative study about long-term outcomes after ESD and gastrectomy. Therefore, this protocol aims to evaluate overall survival rate, tumor recurrence, development of metachronous cancers between ESD and surgery groups.

ELIGIBILITY:
Inclusion Criteria:

* differentiated type mucosal cancer without ulceration, regardless of tumor size
* differentiated type mucosal cancer with ulceration ≤ 3 cm in diameter
* superficial (SM1 < 500 μm) submucosal cancer ≤ 3 cm in diameter
* undifferentiated type mucosal cancer without ulceration ≤ 2 cm in diameter

Exclusion Criteria:

* early gastric cancer in a remnant stomach
* gastrectomy due to metachronous lesions during follow-up period
* post-ESD additional surgery due to high risk of lymph node metastasis or the possibility of residual tumor

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with early gastric cancer were treated by surgery or ESD at a single, tertiary-care, academic medical center.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2003-05; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Patient's death | up to 5 years

SECONDARY OUTCOMES:
Tumor recurrence | up to 5 years
Development of metachronous cancers | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Cho, M.D., Principal Investigator — Soonchunhyang University Hospital, Seoul, Korea
Locations (1):
- Soonchunhyang University Hospital, Seoul, South Korea